CLINICAL TRIAL: NCT03191097
Title: Randomised Double-blind Placebo Controlled Multicenter Clinical Trial of Efficacy and Safety of Ingavirin® Capsules 30mg, in Daily Dose 60mg for the Treatment of Influenza and Other Acute Respiratory Viral Infections at Children 7-12 y.o.
Brief Title: Efficacy and Safety Study of Ingavirin® to Treat Influenza and Acute Respiratory Viral Infections in Children 7-12 y.o.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Collaborators: Atlant Clinical Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4K/2013
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Influenza, Human; Acute Respiratory Infection; Viral Infection; Common Cold
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Common Cold | interventions — pentanedioic acid imidazolyl ethanamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ingavirin (Experimental)
  Interventions: Drug: Ingavirin
- Placebo oral capsule (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Ingavirin — Ingavirin capsules 60 mg once daily, regardless of meal, for 5 days.
  Other Names: Imidazolyl ethanamide pentandioic acid
  Arms: Ingavirin
Drug: Placebo oral capsule — Placebo, capsules daily for 5 days.
  Arms: Placebo oral capsule

SUMMARY:
The purpose of this study is to determine whether Ingavirin ® dosed 60 mg daily is effective and safe in the treatment of influenza and other acute respiratory viral infections in 7-12 years old patients.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent form signed by the patient's parent/adoptive parent to participate in the clinical study
* Male and female patients aged 7-12
* Patients with moderate course of influenza or other acute respiratory viral infections (AVRI)
* Patients with clinically diagnosed influenza or other ARVI based on the body temperature > 37,5 ° C, not less than 1 of the following other symptoms of intoxication and not less than 1 of the following of catarrhal symptoms:
* Intoxication symptoms: headache, malaise, myalgia, pain in the eyeballs;
* Catarrhal symptoms: sore throat, rhinorrhea, cough, nasal congestion
* Uncomplicated course of influenza and other ARVI
* Interval between onset of symptoms and enrollment to the study of not more than 36 hours

Exclusion Criteria:

* Complicated course of influenza and other acute respiratory viral infections
* Treatment with antiviral drugs (antivirals, interferons and interferon inducers), drugs with immunomodulatory effects or antibiotics with systemic and local action within 7 days prior to the screening visit
* Severe influenza or other ARVI with symptoms of cardiovascular disease, and other symptoms of infectious-toxic shock, and meningoencephalitic syndromes
* Signs of primary viral pneumonia development (presence of two or more of the following symptoms): shortness of breath, chest pain when coughing, systemic cyanosis, dullness of percussion sound at symmetrical assessment of the upper and lower parts of the lungs
* Infectious diseases within the last week prior to enrollment
* "RRI children" (incidence of ARVI within the last 12 months is 6 times or more)
* Asthma history
* History of increased seizure activity
* Severe decompensated or unstable medical or psychiatric conditions (any diseases or conditions that threaten the life of the patient or worsen the patient's prognosis and also make it impossible to conduct a clinical study in the patient).
* Cancer, HIV infection, tuberculosis, including those in history
* Hypersensitivity to imidazolyl ethanamide pentandioic acid and/or excipients of Ingavirin product
* Diabetes, lactose intolerance, lactase deficiency, glucose-galactose malabsorption, deficiency of sucrase/isomaltase, fructose intolerance, hereditary glucose malabsorption, deficiency of glucose-6-phosphate dehydrogenase
* Participation of the patient in any other clinical trial within the last 90 days prior to enrollment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time to resolution of fever | 7 ± 1 days
  Time from the start of study treatment to resolution of fever ( t ≤ 36,9 ºС)

SECONDARY OUTCOMES:
Time to resolution of intoxication symptoms | 7 ± 1 days
  Time from the start of study treatment to resolution of all intoxication symptoms.
Time to resolution of catarrhal symptoms | 7 ± 1 days
  Time from the start of study treatment to resolution of all catarrhal symptoms.

OTHER OUTCOMES:
Proportion of subjects with resolution of fever | 7 ± 1
  Proportion of subjects with resolution of fever by 1st, 2nd, 3rd, 4th and 5th days of treatment
Proportion of subjects with development of complications of Influenza or other acute respiratory viral infection | 21 ± 1
  Proportion of subjects who developed complications during treatment period (7 ± 1 days) and follow-up period (21 ± 1 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Zakharova, MD, PhD, Study Director — Valenta Pharm JSC
Locations (11):
- Russia (11):
  - GBOU VPO "Kazan State Medical University" of Ministry of Health of Russian Federation, Kazan'
  - Krasnoyarsk State Medical University named after Prof. V.F.Voino-Yasenetsky, Krasnoyarsk
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Novosibirsk State Medical University, Novosibirsk
  - City Pediatric Outpatient Clinic number 5, Perm
  - Rostov State Medical University, Rostov-on-Don
  - Pediatrics outpatient clinic number 4 of Rostov-na-Donu, Rostov-on-Don
  - Ogarev Mordovia State University, Saransk
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - GBOU VPO "Yaroslavl State Medical University" of Ministry of Health of Russian Federation, Yaroslavl
  - Pediatrician City Hospital number 11, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] I.M. Farber, N.A. Geppe, D.V. Reikhart, V.E. Nebolsin, V.S. Arnautov, A.A. Globenko. Therapy for influenza and acute respiratory viral infection in young and middle-aged schoolchildren: Effect of Ingavirin® on intoxication, fever, and catarrhal syndromes. Ros Vestn Perinatol Pediat 2016; 2:115-120. Russian.
- [Result] N.A. Geppe, E.D. Teplyakova, A.A. Shuldyakov, E.P. Lyapina, O.A. Perminova, G.P. Martynova, I.G. Sitnikov, V.A. Anohin, G.R. Fatkullina, V.V. Romanenko, A.A. Savisko, E.G. Kondyurina, L.A. Balykova. Innovations in pediatrics: the optimal clinical effect In acute respiratory viral infections treatment In children with complex action drug. Pediatry 2016, 2(95), 97-103. Russian.